CLINICAL TRIAL: NCT06556316
Title: The Brain Injury Neurorehabilitation Project
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Fofi Constantinidou, Professor of Psychology, University of Cyprus
Other Study IDs: Excellence/1216/0411; Excellence/0918/0117 (Other Grant/Funding Number: Research and Innovation Foundation)
Record Dates: First submitted 2024-07-30; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Traumatic Brain Injury; CVA (Cerebrovascular Accident)
Keywords: ABI; CVA; Cognition; Psychosocial; Quality of life; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Patients with Moderate to Severe TBI who will receive cognitive rehabilitation: Adults with a history of moderate to severe TBI who will receive cognitive rehabilitation through the Categorization Program, a hierarchical remedial intervention
  Interventions: Behavioral: Cognitive Intervention with the Categorization Program
- Patients with Moderate to Severe TBI who will receive psychosocial intervention: Adults with a history of moderate to severe TBI who will receive group intervention via the Social Cognitive Communication Program (SocCom)
  Interventions: Behavioral: Social Cognitive Communication Program
- Patients with a history of CVA who will receive psychosocial intervention: Adults with a history of CVA (hemorrhagic or ischemic) who will receive group intervention via the Social Cognitive Communication Program (SocCom)
  Interventions: Behavioral: Social Cognitive Communication Program
- Patients with a history of CVA who will receive psychosocial intervention and tDCS: Adults with a history of CVA (hemorrhagic or ischemic) who will receive group intervention via the Social Cognitive Communication Program (SocCom) and tDCS treatment
  Interventions: Behavioral: Social Cognitive Communication Program; Device: Non-Invasive Brain Stimulation with tDCS
- Patients with TBI who will receive psychosocial intervention & TDCS: Adults with a history of moderate to severe TBI who will receive group intervention via the Social Cognitive Communication Program (SocCom) and tDCS treatment
  Interventions: Behavioral: Social Cognitive Communication Program; Device: Non-Invasive Brain Stimulation with tDCS
- Patients with TBI receiving group psychosocial intervention and the Categorization Program: Adults with a history of moderate to severe TBI who will receive cognitive rehabilitation through the CP and group intervention with the SocCom treatment
  Interventions: Behavioral: Cognitive Intervention with the Categorization Program; Behavioral: Social Cognitive Communication Program

INTERVENTIONS:
Behavioral: Cognitive Intervention with the Categorization Program — Cognitive intervention delivered individually. This is a hierarchical cognitive rehabilitation program
  Other Names: CP
  Groups: Patients with Moderate to Severe TBI who will receive cognitive rehabilitation; Patients with TBI receiving group psychosocial intervention and the Categorization Program
Behavioral: Social Cognitive Communication Program — An 11 week group intervention targeting social and cognitive-communication abilities
  Other Names: Soc Com
  Groups: Patients with Moderate to Severe TBI who will receive psychosocial intervention; Patients with TBI receiving group psychosocial intervention and the Categorization Program; Patients with TBI who will receive psychosocial intervention & TDCS; Patients with a history of CVA who will receive psychosocial intervention; Patients with a history of CVA who will receive psychosocial intervention and tDCS
Device: Non-Invasive Brain Stimulation with tDCS — 20 minute tDCS intervention as a non-invasive neuromodulation treatment
  Other Names: tDCS Intervention
  Groups: Patients with TBI who will receive psychosocial intervention & TDCS; Patients with a history of CVA who will receive psychosocial intervention and tDCS

SUMMARY:
The primary objective of The Brain Injury Neurorehabilitation Project is a systematic effort to generate cutting edge research in brain injury and cognitive rehabilitation that will advance neurorehabilitation research. It will establish the first surveillance system and implement multimodal data to characterize the long-term effects of moderate to severe TBI. Additionally, the project will implement innovative rehabilitation methodologies, namely, cognitive training, social communication deficits and non-invasive brain stimulation with tDCS, to determine which modality can improve neurocognitive and psychosocial performance in adult ABI. Two funded projects, BRAIN-REHAB & ACESO are incorporated in this project.

DETAILED DESCRIPTION:
Acquired Brain Injury resulting from a TBI or CVA is a primary cause of chronic disability and unemployment, resulting in significant health, societal, and financial burden. The Brain Injury Neurorehabilitation Project is part of a systematic effort to study ABI in Cyprus. It is an umbrella project designed to generate cutting edge research in brain injury and cognitive rehabilitation that will advance neurorehabilitation research. Patients with TBI and strokes are often faced with cognitive and behavioral difficulties that interfere with their ability to return to productive living, thus contributing to unemployment, social isolation and low quality of life for decades post injury. The scientific objectives will address the aforementioned challenge. First, the project will establish the first TBI surveillance system in Cyprus and implement epidemiologically-principled and systematic data collection from large cohorts across the severity continuum. It will integrate neuropsychological, lifestyle, injury, imaging, genetic, and biological data using state of the art computational methods and quantitatively assess the exact contribution of critical variables to brain injury recovery. Second, the project will determine the effectiveness of a theory-driven neurocognitive therapy program, the Categorization Program (CP) in combination with a social-communication training during the chronic phase of the recovery process. It is hypothesized that the combination of remedial cognitive and social-communication training will yield improvement in functioning with sustainable long term effects. Additionally, the project will implement non-invasive brain stimulation (NIBS) in combination with the social-communication intervention to determine the utility of NIBS and specifically tDCS, in improving cognitive performance and psychosocial functioning. Through innovative research and development of new methods and technologies, the project will advance the State-of-the-Art by producing cutting edge research with international impact while contributing to the development of personalized medicine and improvement of rehabilitation outcomes and reduction of disability in Cyprus.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe TBI or hospitalization due to CVA

Exclusion Criteria:

* history of neurodevelopmental disorder, prior neurological history or psychiatric history requiring hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survivors of ABI (TBI and CVA) who have been hospitalized and are at the chronic phases of their condition. They will be recruited from rehabilitation centers, patient advocacy groups and the major trauma hospital in Cyprus.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Memory | Administered pre & post training at 3 & 6 months follow up
  The Greek version of the Auditory Verbal Learning Test will be used as a key outcome for memory. The test consists of a list of 15 items read to the participant, and the participant is required to recall as many items from the list. Maximum score per trial is 15. The process is repeated 5 times (presentation of the list and subsequent recall) for a possible maximum score of 60. A thirty-minute delay is also included after the five learning trials. The measure allows exploring a number of memory processes, such as short term memory (trial one), working memory (list learning across the five trials) and episodic memory (ability to recall items on the list after the 30-minute delay).
Language | Administered Pre and Post training at 3 & 6 months follow up
  Expressive and receptive language, including naming and verbal fluency, will be used. For this task, we will use the Greek short version of the Peabody Picture Vocabulary test (maximum score of 32) the Greek Short Version of the Boston Naming Test (maximum score of 20). In addition, animal naming in 60 seconds and words from letter F in 60 seconds will be used for verbal fluency. For all tasks, higher scores indicate better performance.
Executive Functioning | Administered pre & post training at 3 & 6 months follow up
  Laboratory and structured questionnaires will be used to assess executive functions. Laboratory tests include the Trail Making A and B (performance is measured in seconds; the faster, the better), and the Symbol Digits Modalities task (completion of as many items as possible in 90 seconds; higher score is better). In addition, the Dysexecutive Questionnaire will be completed by the participant and a close informant, to assess everyday executive functioning abilities. Maximum score is 148 and the lower score indicates better executive abilities.

SECONDARY OUTCOMES:
WHO-BREF Quality of Life | Adminsitered pre & post training at 3 & 6 months follow up
  This measure by the World Health Organization is a widely used measure of general quality of life across key domains: Psychological Health, Physical Health, Environment/Support. Higher scores indicate better quality of life. There is no specific cut-off score. Statements are rated on a likert scale. Higher scores indicate greater satisfaction with one's quality of life.
Depression | Adminisered pre & post training at 3 & 6 months follow up
  The Greek version of the Beck Depression Inventory will be used. Higher scores indicate greater levels of depressive symptomatology. The score of 15 and higher indicates mild levels of depression. Maximum score is 63.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided
Certain aspects of the study protocol may be shared after publication of study results